CLINICAL TRIAL: NCT03446664
Title: Microburst VNS Therapy Feasibility Study in Subjects With Refractory Epilepsy
Brief Title: Microburst Vagus Nerve Stimulator (VNS) Therapy Feasibility Study
Acronym: Microburst
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LNN001
Record Dates: First submitted 2018-02-09; First posted 2018-02-27 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Epilepsies, Partial; Epilepsy, Tonic-Clonic
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy, Tonic-Clonic

STUDY DESIGN:
Intervention Model Description: Two cohorts of subjects with refractory epilepsy; (1) subjects with primary generalized tonic-clonic seizures and (2) subjects with partial onset seizures including complex partial seizures with or without secondary generalization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Microburst Stimulation (Experimental): Microburst stimulation to tolerability and effectiveness
  Interventions: Device: Microburst Stimulation

INTERVENTIONS:
Device: Microburst Stimulation — Implantable generator with new stimulation feature under study to determine the safety and effectiveness of device stimulation on different seizure types.

SUMMARY:
Evaluate the initial safety and effectiveness of Microburst VNS stimulation in subjects with refractory epilepsy.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of medically refractory epilepsy with primary generalized tonic-clonic seizures (limited to 20 subjects) or partial onset seizures including complex partial seizures with or without secondary generalization (limited to 20 subjects).
2. Must be on adjunctive antiepileptic medications.
3. Willing and capable to undergo multiple evaluations with functional magnetic resonance imaging (fMRI), electroencephalogram (EEG) and electrocardiogram (ECG).

4(A) For subjects with partial onset seizures: An average of ≥ 3 countable seizures per month based on seizure diary during the 3 month baseline period and no seizure-free interval greater than 30 days during those 3 months.

4(B) For subjects with PGTCs: Have at least ≥ 3 countable seizures during the 3 month baseline period. Note: Each seizure within a cluster may be counted as separate seizures.

5. 12 years of age or older.

6. Subject is a male or non-pregnant female adequately protected from conception. Females of childbearing potential must use an acceptable method of birth control.

7. Provide written informed consent-assent/Health Insurance Portability and Accountability Act (HIPAA) authorization and self-reported measures with minimal assistance as determined by the investigator.

Exclusion Criteria:

1. Currently using, or are expected to use, short-wave diathermy, microwave diathermy, or therapeutic ultrasound diathermy.
2. A VNS Therapy System implant would (in the investigator's judgment) pose an unacceptable surgical or medical risk for the subject.
3. A planned procedure that is contraindicated for VNS therapy.
4. History of implantation of the VNS Therapy System.
5. Currently receiving treatment from an active implantable medical device.
6. Presence of contraindications to MRI per the MRI subject screening record.
7. Known clinically meaningful cardiovascular arrhythmias currently being managed by devices or treatments that interfere with normal intrinsic heart rate responses (e.g., pacemaker dependency, implantable defibrillator, beta adrenergic blocker medications).
8. History of chronotropic incompetence (commonly seen in subjects with sustained bradycardia [heart rate < 50 bpm]).
9. Cognitive or psychiatric deficit that in the investigator's judgment would interfere with the subject's ability to accurately complete study assessments.
10. History of status epilepticus within 1 year of study enrollment.
11. Dependent on alcohol or narcotic drugs as defined by DSM IV-TR within the past 2 years, based on history. Tests for drug or alcohol use will not be administered.
12. Currently being treated with prescribed medication that contains cannabis or cannabis related substance including recreational use.
13. Any history of psychogenic non-epileptic seizures.
14. Currently participating in another clinical study without LivaNova written approval.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Efficacy Primary Endpoint: Percent change from baseline in seizure frequency | Up to 12 months study visit
  For the primary endpoint, the change in the seizure frequency per month compared to baseline will be evaluated for each subject at follow-up visits month 6 and 12.
Safety Primary Endpoint: Occurrence of stimulation related Adverse Events | Up to 12 months study visit
  Assess stimulation/device related adverse events at follow-up visits month 6 and 12.

SECONDARY OUTCOMES:
Change from baseline in seizure frequency per month based on seizure diary provided by the sponsor | Up to 12 months study visit
Change from baseline in seizure severity | Up to 12 months study visit
  As measured by the Seizure Severity Questionnaire (SSQ) scale (Cramer, 2002).
Change from baseline in quality of life | Up to 12 months study visit
  As measured by the QOLIE-31-P for adults 18 years and older (Cramer et al.; 1998) and QOLIE-AD-48 for adolescents 12 to 17 years (Cramer et al.; 1999).
Change from baseline in antiepileptic drug (AED) load | Up to 12 months study visit
  Estimated as the sum of the prescribed daily dose (PDD)/defined daily dose (DDD) ratios for each AED included in the treatment regimen (Deckers et al., 1997), where DDD (WHO ATC/DDD index) corresponds to the assumed average therapeutic daily dose of a drug used for its main indication.
Suicidality as measured by the Columbia Suicide Severity Rating Scale (C-SSRS) | Up to 12 months study visit
All adverse events | Up to 12 months visit

CONTACTS AND LOCATIONS:
Overall Officials: Selim Benbadis, MD, Principal Investigator — University of South Florida Health
Locations (9):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Denver Colorado, Denver, Colorado
  - Mayo Clinic Florida, Jacksonville, Florida
  - Rush University, Chicago, Illinois
  - Northwestern University, Evanston, Illinois
  - Weil-Cornell Medical College, Ithaca, New York
  - Duke University, Durham, North Carolina
  - University of Utah, Salt Lake City, Utah
- Ghent University Hosptial, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Szaflarski JP, Allendorfer JB, Begnaud J, Ranuzzi G, Shamshiri E, Verner R; Microburst Study Group. Optimized microburst VNS elicits fMRI responses beyond thalamic-specific response from standard VNS. Ann Clin Transl Neurol. 2024 May;11(5):1135-1147. doi: 10.1002/acn3.52029. Epub 2024 Mar 26. PMID 38532258
- [Derived] Drees C, Afra P, Verner R, Kaye L, Keith A, Jiang M, Szaflarski JP, Nichol K; Microburst Study Group. Feasibility study of microburst VNS therapy in drug-resistant focal and generalized epilepsy. Brain Stimul. 2024 Mar-Apr;17(2):382-391. doi: 10.1016/j.brs.2024.03.010. Epub 2024 Mar 16. PMID 38499287
- [Derived] Verner R, Szaflarski JP, Allendorfer JB, Vonck K, Giannicola G; Microburst Study Group. Modulation of the thalamus by microburst vagus nerve stimulation: a feasibility study protocol. Front Neurol. 2023 Jun 13;14:1169161. doi: 10.3389/fneur.2023.1169161. eCollection 2023. PMID 37384278